CLINICAL TRIAL: NCT00036933
Title: Vaccination Of Prostate Cancer Patients With A Bivalent Vaccine Containing MUC-2 Glycopeptide And Globo H Conjugates Plus The Immunological Adjuvant QS21
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-140; P30CA008748 (NIH); MSKCC-01140; NCI-G02-2064
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — saponin QA-21V1

ARMS (1):
- vaccine (Experimental): Patients receive glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant QS21 subcutaneously once weekly on weeks 0-2, 6, 14, and 26 in the absence of unacceptable toxicity. Patients whose antibody titers against Globo-H or MUC-2 antigens fall below 1/40 and who have no disease progression may receive a seventh vaccination after week 50.
  Patients are followed every 3 months for 1 year or until biochemical relapse or radiographic disease progression.
  Interventions: Biological: MUC-2-Globo H-KLH conjugate vaccine; Biological: QS21

INTERVENTIONS:
Biological: MUC-2-Globo H-KLH conjugate vaccine
Biological: QS21

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Biological therapies such as QS21 use different ways to stimulate the immune system and stop cancer cells from growing. Combining vaccine therapy with QS21 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy with QS21 in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant QS21 in patients with prostate cancer.
* Determine the antibody response in patients treated with this vaccination therapy.
* Assess post-immunization changes in PSA levels and other objective parameters of disease (radionuclide bone scan) in patients treated with this vaccination therapy.

OUTLINE: Patients receive glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant QS21 subcutaneously once weekly on weeks 0-2, 6, 14, and 26 in the absence of unacceptable toxicity. Patients whose antibody titers against Globo-H or MUC-2 antigens fall below 1/40 and who have no disease progression may receive a seventh vaccination after week 50.

Patients are followed every 3 months for 1 year or until biochemical relapse or radiographic disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Disease progression after primary surgery (radical prostatectomy) or radiotherapy with or without prior neoadjuvant androgen ablation

  * Minimum of 3 rising PSA values, taken at least 2 weeks apart, with more than a 50% rise in PSA level above the baseline value (1.0 ng/mL post -prostatectomy or 2.0 ng/mL post-radiotherapy)
  * Received prior intermittent hormonal therapy after prior primary therapy
  * Non-castrate levels of testosterone (more than 50 ng/mL)
* Evaluable disease (by serial changes in PSA)
* No radiographic evidence of metastatic disease
* No active CNS or epidural tumor
* No soft tissue and/or bone disease
* No androgen-independence with no evidence of radiographic disease
* May not be symptomatic or anticipated to develop symptoms within 6 months of study entry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT less than 3 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 40 mL/min

Cardiovascular:

* No clinically significant cardiac disease (New York Heart Association class III or IV)

Pulmonary:

* No severe debilitating pulmonary disease

Other:

* No allergy to seafood (shellfish)
* No other active malignancy within the past 5 years except nonmelanoma skin cancer
* No infection requiring antibiotics
* No narcotic-dependent pain
* No positive stool guaiac unless associated with hemorrhoids or prior documented radiation-induced proctitis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* See Chemotherapy
* At least 2 weeks since change in hormonal therapy (e.g., prednisone or dexamethasone) except to maintain castrate levels of testosterone

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent irradiation of only measurable lesion

Surgery:

* See Disease Characteristics
* No concurrent surgery of only measurable lesion

Other:

* Recovered from prior therapy
* At least 8 weeks since prior suramin and/or documented plasma concentration of suramin if less than 50 micrograms/mL (replacement hydrocortisone allowed)
* No other concurrent oncolytic agents
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
safety | 2 years

SECONDARY OUTCOMES:
response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States